CLINICAL TRIAL: NCT05988983
Title: The Over The Counter Pill National Study
Status: Active, not recruiting | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Collaborators: Arnold Ventures (Unknown)
Responsible Party: Principal Investigator, Maria Rodriguez, MD, MPH, Professor of Obstetrics and Gynecology, Oregon Health and Science University
Other Study IDs: OHSU IRB 25984
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-04

CONDITIONS: Contraception; Contraception Behavior; Contraceptive Usage; Health Care Utilization
MeSH Terms: conditions — Contraception Behavior; Patient Acceptance of Health Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- OTC users: Participants using the oral contraceptive pill purchased over the counter
  Interventions: Other: Availability of OTC contraceptive pill
- Rx users: Participants using the oral contraceptive pill received by a prescription

INTERVENTIONS:
Other: Availability of OTC contraceptive pill — Over the counter contraceptive pill
  Groups: OTC users

SUMMARY:
This is a prospective cohort study of individuals purchasing the oral contraceptive pill over the counter (OTC) in pharmacies in 32 US states. The comparison group is people receiving a prescription (Rx) for oral contraception. Both groups will be followed for one year to examine contraceptive continuation rates. This study will also identify who is using the pill OTC and why and evaluate differences in pregnancy intention and measures of contraceptive agency between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Capable of pregnancy
* Purchasing oral contraception at a participating pharmacy

Exclusion Criteria:

* Using the pill for non contraceptive indications

Ages: 12 Years to 51 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Individuals aged 12 to 51 who are obtaining the oral contraceptive pill at a pharmacy for the purposes of pregnancy prevention.
Sampling Method: Probability Sample
Enrollment: 1026 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
12 month contraceptive continuation rates | 12 months
  Difference in proportion of participants using contraception 12 months after starting between over the counter and prescription groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Undecided